CLINICAL TRIAL: NCT01543529
Title: A Single Center, Randomized, Double-blind, Single-dose, Four Period, Crossover Study to Investigate Pharmacodynamics and Pharmacokinetics of RO4917838 Alone or With Concomitant Administration of Alcohol in Healthy Volunteers
Brief Title: A Pharmacodynamic and Pharmacokinetic Study of RO4917838 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BP28180
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- RO4917838 + non-alcoholic drink (Active Comparator)
  Interventions: Drug: RO4917838
- RO4917838 + alcohol (Experimental)
  Interventions: Drug: RO4917838; Other: Alcohol
- RO4917838 placebo + alcohol (Placebo Comparator)
  Interventions: Drug: Placebo to RO4917838; Other: Alcohol
- RO4917838 placebo + non-alcoholic drink (Placebo Comparator)
  Interventions: Drug: Placebo to RO4917838

INTERVENTIONS:
Drug: RO4917838 — Single dose of RO4917838
  Arms: RO4917838 + alcohol; RO4917838 + non-alcoholic drink
Drug: Placebo to RO4917838 — Single dose of placebo to RO4917838
  Arms: RO4917838 placebo + alcohol; RO4917838 placebo + non-alcoholic drink
Other: Alcohol — Standard alcoholic drink
  Arms: RO4917838 + alcohol; RO4917838 placebo + alcohol

SUMMARY:
This single-center, randomized, double-blind, four-period crossover study will investigate the effect of alcohol on the pharmacodynamics and pharmacokinetics of RO4917838 in healthy volunteers. Healthy volunteers will receive 4 treatments in a randomized order: single dose of RO4917838 and alcohol, RO4917838 and non-alcoholic drink, placebo to RO4917838 and alcohol, and placebo to RO4917838 and non-alcoholic drink.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, 18 to 45 years, inclusive
* Body Mass Index (BMI) 18 to 30 kg/m2, inclusive
* Non-smoker or smoker of fewer than 10 cigarettes per day
* Females, who are not menopausal must agree to use two adequate methods of contraception

Exclusion Criteria:

* Any current medical condition or disease that would render the volunteer unsuitable for the study, or would place the volunteer at undue risk
* History of alcoholism
* History of drug abuse and/or addiction within one year of study start
* History of any significant disease (e.g., cardiovascular, hepatic, renal) or cancer

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2012-06-04 (Actual); Study Completion 2012-06-04 (Actual)

PRIMARY OUTCOMES:
Effect of alcohol on pharmacodynamics (Cognitive test battery) of RO4917838 | Day 1 of each treatment period

SECONDARY OUTCOMES:
Effect of alcohol on pharmacokinetics (Area under the concentration time curve) of RO4917838 | Days 1, 2, 3, 4, 6, and 8 of each treatment period
Safety: Incidence of adverse events | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- BIOTRIAL, Rennes, France